CLINICAL TRIAL: NCT05677373
Title: Phase I/II Study of BET and MEK Inhibition in Advanced Uveal Melanoma
Brief Title: Testing the Safety and Effectiveness of Combining Two Drugs, PLX2853 and Trametinib in the Treatment of Advanced Uveal Melanoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The drug company supporting this trial has withdrawn support, including the ability to provide study agent.
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A092106
Record Dates: First submitted 2023-01-09; First posted 2023-01-10 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Advanced Uveal Melanoma; Metastatic Uveal Melanoma; Unresectable Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — trametinib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (PLX2853, trametinib) (Experimental): Patients receive PLX2853 PO in combination with trametinib PO throughout the study. Patients also undergo collection of blood at screening and on study. Patients also undergo CT or MRI with contrast and collection of blood at screening and on study.
  Interventions: Drug: BRD4 Inhibitor PLX2853; Drug: Trametinib; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen collection

INTERVENTIONS:
Drug: BRD4 Inhibitor PLX2853 — Given PO
  Other Names: PLX 2853; PLX-2853; PLX2853
Drug: Trametinib — Given PO
  Other Names: 871700-17-3; GSK1120212; JTP-74057
Procedure: Computed Tomography — Undergo CT with contrast
  Other Names: CAT; CAT scan; Computed Axial Tomography; CT Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI with contrast
  Other Names: MRI
Procedure: Biospecimen collection — Undergo collection of blood
Procedure: Biospecimen collection — Correlative studies

SUMMARY:
This phase I/II trial tests the safety, side effects, and best dose of PLX2853 in combination with trametinib in treating patients with uveal (eye) melanoma that has spread to other places in the body (metastatic) or nearby tissues or lymph nodes (locally advanced), or that cannot be removed by surgery (unresectable). PLX2853 works by targeting and inhibiting certain activities within cells that promote tumor growth. By inhibiting these activities, PLX2853 may help to stabilize or reduce the growth of tumor cells. Trametinib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals tumor cells to multiply. This helps stop the spread of tumor cells. Giving PLX2853 in combination with trametinib may help to shrink and stabilize tumor cells in patients with advanced uveal melanoma.

DETAILED DESCRIPTION:
CO-PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose(s) (MTD(s)) and recommended phase II dose. (Phase I) II. To evaluate whether combination BRD4 inhibitor PLX2853 (PLX2853) and trametinib demonstrate clinical activity in advanced uveal melanoma (UM), as determined by a best response rate of 25% compared to a historical rate of 10%. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate (ORR) associated with combination PLX2853 and trametinib.

II. To evaluate the progression-free survival (PFS) associated with combination PLX2853 and trametinib.

III. To evaluate the overall survival (OS) associated with combination PLX2853 and trametinib.

IV. To characterize the adverse event profile associated with combination PLX2853 and trametinib.

PHARMACOKINETICS SECONDARY OBJECTIVE:

I. To evaluate the pharmacokinetic profile of combination PLX2853 and trametinib.

OUTLINE: This is a phase I dose-escalation study of PLX2853 and trametinib followed by a phase II study.

Patients receive PLX2853 orally (PO) in combination with trametinib PO throughout the study. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) with contrast and collection of blood at screening and on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented advanced uveal melanoma. Pathology review and confirmation of diagnosis will occur at the site enrolling the patient on this study. Patients must have locally advanced unresectable or metastatic uveal melanoma (UM).
* Patients must have at least one lesion which is measurable according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria. Measurable disease is not required in the phase I portion
* Patients may be treatment-naïve or have received any number of prior systemic or liver-directed therapies for advanced UM. There are no maximum number of prior therapies received
* There is no specified washout time for prior therapies however patients must have fully recovered from acute toxicities related to prior anti-cancer therapies including

  * Cytotoxic therapies, immunotherapy, small molecule targeted agents, cell therapy, liver-directed therapy, or radiation therapy
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown. Therefore, for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Hemoglobin >= 9g/dL (transfusions to achieve this level are allowed)
* Platelet count >= 100,000/mm^3
* Creatinine clearance >= 45 mL/minute (per Cockcroft-Gault equation)
* Total bilirubin =<1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) =< 3 x upper limit of normal (ULN)
* Prothrombin time (PT)/international normalized ratio (INR) =< 1.5 x upper limit of normal (ULN)
* No history of any medical condition such as uncontrolled infection (including hepatitis B [HepB], hepatitis C [HepC]), uncontrolled diabetes mellitus or cardiac disease which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient
* Patients who are human immunodeficiency virus (HIV)-infected on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible
* Patients with a new or progressive brain metastases (active brain metastases) or leptomeningeal disease if the treating physician determines that immediate central nervous system (CNS) specific treatment is not required and is unlikely to be required during the first cycle of therapy are eligible
* Patients with a known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification with a class 2B or better are eligible
* Patients must be able to obtain confirmation of payment coverage (insurance or other) for trametinib * Trametinib will not be provided by the Alliance and must be obtained through commercial or other mechanisms independent of the clinical trial. Confirmation of payment coverage or medication access must be obtained by treating physician prior to registration

Exclusion Criteria

* Patients must not have received prior treatment with a BET or MEK inhibitor
* No patients who cannot swallow oral formulations of the agent(s)
* Chronic concomitant treatment with strong inhibitors of CYP3A4 is not allowed on this study. Patients on strong CYP3A4 inhibitors must discontinue the drug for 14 days prior to registration on the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-13 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Phase I) | Up to 28 days (Cycle 1)
Recommended Phase 2 Dose (RP2D) (Phase I) | Up to 28 days (Cycle 1)
  Will be found using a Keyboard design which will be the dose with an estimated dose-limiting toxicity (DLT) rate closest to 25% (the target DLT rate).

SECONDARY OUTCOMES:
Overall response rate (ORR) (phase II) | 2 years
  Defined as the number of patients that achieve a best response of PR or better divided by the total number of evaluable patients. Will be evaluated using a Simon two-stage mini-max design using a historical response rate of 10% based on some prior work in this disease population with chemotherapy and targeted therapy. A 95% confidence interval for this estimate will also be calculated based on properties of the binomial distribution.
Median progression-free survival (PFS) | At 1 year
  The Kaplan-Meier (KM) method will be used to estimate the median PFS time. A 95% confidence interval for the median PFS time will also be calculated using KM methodology.
Progression free survival (PFS) | From registration until first evidence of progression (or death), assessed up to 2 years
  Will be estimated using Kaplan-Meier method, and a 95% confidence interval will also be calculated using KM methodology.
Median overall survival (OS) | At 1 year
  The Kaplan-Meier method will be used to estimate the median PFS time. A 95% confidence interval for the median PFS time will also be calculated using KM methodology.
Overall survival (OS) | From registration until death due to any cause, assessed up to 2 years
  Will be estimated using Kaplan-Meier method, and a 95% confidence interval will also be calculated using KM methodology.
Incidence of adverse events | Up to 2 years
  Adverse events will be recorded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 for each patient. Frequency tables and summary statistics will be used and with the appropriate methods of evaluating categorical and continuous data.
Systemic exposure to trametinib and PLX2853 - pharmacokinetics | Up to 2 years
  Systemic exposure to trametinib and PLX2853 will be assessed by determining trough plasma concentrations (Ctrough, Cmin), which is the concentration in a sample collected immediately prior to a next dose. Ctrough will be determined throughout the first two treatment cycles on day 1 and day 15. Ctrough of trametinib and PLX2853 will be summarized using descriptive statistics. Dose dependency of Ctrough in phase 1 will be investigated using exploratory statistics. Potential changes in systemic exposure to either trametinib and/or PLX2853 over time will be explored by investigating changes in Ctrough during the two cycles. In addition, will use population PK models combined with the Ctroughs to describe the full PK of trametinib and PLX2853.

IPD SHARING:
Plan to Share IPD: Undecided